CLINICAL TRIAL: NCT05802108
Title: Effect of PCSK9 Inhibitor on Retinal Microvessels in Patients With Coronary Heart Disease After Intensive Lipid-lowering Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zibo Central Hospital (Other Government)
Responsible Party: Principal Investigator, Bo Li, Clinical Professor；Department of Cardiology, Zibo Central Hospital, Zibo Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZiboCH2
Record Dates: First submitted 2023-03-11; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Adverse Effect of Cardiovascular Medications (Diagnosis)
MeSH Terms: conditions — Disease | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): evolocumab combined with statins
  Interventions: Drug: Evolocumab combined with statins
- Control Group (Other): statins only
  Interventions: Drug: Statin

INTERVENTIONS:
Drug: Evolocumab combined with statins — The experimental group was treated with evolocumab combined with statin for lipid-lowering
  Other Names: drug1
  Arms: Experimental Group
Drug: Statin — the control group was treated with statin only for lipid-lowering
  Other Names: drug2
  Arms: Control Group

SUMMARY:
In patients with coronary heart disease who were treated with PCSK9 inhibitor evolocumab for intensive lipid-lowering therapy, the changes of retinal microvessels were measured with OCTA (Optical Coherence Tomography Angiography)before and after the treatment. The specific indicators included retinal microvessel diameter, macular area，optic disc vascular density and FAZ(Foveal Avascular Zone)area, etc., to clarify the effect of evolocumab on retinal microvessels after intensive lipid-lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-75 years old, gender unlimited;
2. Diagnosed as coronary atherosclerotic heart disease
3. The informed consent for the study has been signed

Exclusion Criteria:

1. Those who are unable to cooperate with the examination;
2. Poor imaging quality of refractive interstitial opacity;
3. Macular edema or complicated with macular membrane and senile macular degeneration;
4. Have a history of previous fundus surgery;
5. Those with eye diseases that can cause changes in the microvessels of the fundus;
6. Abnormal elevated intraocular pressure;
7. Moderate or above refractive error (≥ ± 3 diopters)
8. People with cognitive impairment, material dependence, and serious mental illness;
9. Those who do not cooperate with follow-up;
10. Those who participate in other clinical trials at the same time

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
the main indicator | Up to 12 months
  Video disc area (4.5 × 4.5 mm2) of the radial capillary network (RPC) around the nipple and the macular area (6 × 6 mm2), superficial retinal vascular plexus (SCP) and deep retinal vascular plexus (DCP).

SECONDARY OUTCOMES:
the secondary indicator | Up to 12 months
  The thickness of the retinal nerve fiber layer (RNFL) near the optic disc, the thickness of the retinal ganglion cell layer in the macular region, the area of the avascular zone (FAZ) in the fovea, the changes of blood lipids, and the changes of the diameter of the retinal branch veins near the optic disc

CONTACTS AND LOCATIONS:
Locations (1):
- Zibo Central Hospital, Zibo, Shandong, China